CLINICAL TRIAL: NCT01019161
Title: A Phase I Open, Non-randomised, Single-centre Study to Assess the Metabolism, Excretion and Pharmacokinetics of AZD1152 and AZD1152 hQPA Following Intravenous Administration of [14C]-AZD1152 in Patients With Acute Myeloid Leukaemia (AML)
Brief Title: An Open Label, Single Centre Mass Balance C14 Study in Patients With Acute Myeloid Leukaemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1531C00012
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2010-10

CONDITIONS: Acute Myeloid Leukaemia
Keywords: Acute Myeloid Leukaemia (AML); AML; AZD1152; Pharmacokinetics
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — 2-((3-((4-((5-(2-((3-fluorophenyl)amino)-2-oxoethyl)-1H-pyrazol-3-yl)amino)quinazolin-7-yl)oxy)propyl)(ethyl)amino)ethyl dihydrogen phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD1152 (Experimental): 100 mg Lyophile 5 mL Diluent
  Interventions: Drug: AZD1152
- C14 AZD1152 (Experimental): AZD1152 radiolabelled IV solution. 1.05 mg/ml will be presented as a 15 ml fill in a 20 ml vial.
  Interventions: Drug: C14 AZD1152

INTERVENTIONS:
Drug: AZD1152 — 100mg Lyophile, 5mL Diluent IV infusion
  Arms: AZD1152
Drug: C14 AZD1152 — radiolabelled IV solution, 1.05 mg/ml presented as 15 ml fill in 20ml vial infusion
  Arms: C14 AZD1152

SUMMARY:
The purpose of the study is to assess how AZD1152 is absorbed or excreted in and out of the body in patients with Acute Myeloid Leukaemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory AML for which no standard therapies are anticipated to result in durable remission. Or, patients with newly diagnosed AML who are not considered to be suitable for standard induction and consolidation chemotherapy
* Ability to stay in hospital for up to 9 days on the [14C] AZD1152 treatment cycle.
* Subjects who have relapsed > 1 year following myeloablative therapy with allogeneic bone marrow or stem cell transplantation may be eligible if they have no or limited evidence of extensive graft-versus-host disease

Exclusion Criteria:

* QTc interval ≥470 ms calculated from a single ECG reading or a mean of 3 ECG readings using Fridericia's or Bazett's correction
* Administration of hydroxyurea to control peripheral blood counts is prohibited within 24 hours prior to first dose of study drug
* Any chemotherapy or radiotherapy within 14 days prior to starting the study (not including palliative radiotherapy at focal sites)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The concentration of total radioactivity, AZD1152 and AZD1152 hQPA in plasma and their ratios, the concentration of total radioactivity in blood and its blood/plasma concentration ratios | Day1-10
The derived plasma and urinary pharmacokinetic parameters for AZD1152 and AZD1152 hQPA The percentage of the [14C] AZD1152 dose recovered in urine, faeces and vomit (if presented), and the percentage of radioactive dose recovered overall. | Day1-10

SECONDARY OUTCOMES:
Adverse events (AEs), serious adverse events (SAEs) and deaths, Discontinuations for tolerability reasons, vital signs (temperature, blood pressure [BP], pulse rate and respiratory rate [RR]) | AEs, SAEs, deaths, discontinuations ongoing to completion and vitals over 22 days - Screening, PD Day 1, Days 3, 6, 9, 14, 22
Electrocardiogram (ECG) parameters | Screening, PD Day 1, Day 4
Clinical chemistry, haematology (including clotting parameters) and urinalysis; physical examination | Chemistry/Heamatology - Screening, PD Day 1, Days 3, 6, 9, 14, 22Urinalysis - Screening, PD Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Mike Dennis, MD, Principal Investigator — The Christie Hospital, UK
Locations (1):
- Research Site, Manchester, United Kingdom